CLINICAL TRIAL: NCT01353950
Title: Costimulatory Molecules as Biomarkers in Cystic Fibrosis
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jeffrey Gold, professor, Oregon Health and Science University
Other Study IDs: IRB00007132
Record Dates: First submitted 2011-05-12; First posted 2011-05-16 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Cystic Fibrosis
Keywords: Costimulatory molecules; Cystic Fibrosis; Biomarkers
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, Serum, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adult Cystic Fibrosis Patients: Adults with Cystic Fibrosis will be followed longitudinally for 2 years

SUMMARY:
The purpose of this study is to investigate the expression of a certain class of molecules, called costimulatory molecules, in humans with Cystic Fibrosis. Cystic Fibrosis is a genetic disorder which renders the lung susceptible to persistent inflammation which, at times, can worsen, resulting in accelerated decline in lung function and eventually death or transplant. Our goal is to determine if the levels of costimulatory markers can be used to predict exacerbation and subsequent lung function decline in subjects with Cystic Fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate

Exclusion Criteria:

* Presence of HIV
* Presence of Lymphoma/Leukemia
* Presence of Lung or other solid organ Transplant
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with Cystic Fibrosis
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2011-07; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon health and Sciences University, Portland, Oregon, United States